CLINICAL TRIAL: NCT01095406
Title: Safety, Feasibility and Efficacy of Ventilation Weaning in Children With a Computerized Protocol: a Pilot Study on S1 Ventilator With Intellivent(Hamilton Medical).
Brief Title: Safety and Feasibility Study of a Mechanical Ventilation Computerized Protocol: Intellivent
Acronym: CloserPed
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Philippe Jouvet, Associate Professor, St. Justine's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUSJ-3011
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Mechanical Ventilation Weaning Phase in Children
Keywords: Weaning; closed loop; mechanical ventilation; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S1 ventilation (Active Comparator): Mechanical ventilation with S1 the thrid hour of ventilation
  Interventions: Device: S1 ventilation
- Servo i ventilation (No Intervention): 1 hour ventilation in pressure support mode with Servo i

INTERVENTIONS:
Device: S1 ventilation — Ventilation with a O2 and CO2 controller
  Other Names: Health Canada approval number: 155350
  Arms: S1 ventilation

SUMMARY:
The present protocol will demonstrate the safety, feasibility and efficacy of a newly computerized protocol integrated into a ventilator: S1 ventilator (Hamilton Medical). During ventilation with S1 ventilator, the respiratory support including oxygenation and CO2 removal parameters are continuously adapted to patient respiratory status using science based rules. The present protocol is designed as a pilot evaluative study where the researchers will evaluate the safety, feasibility and efficacy of ventilating children during the weaning phase with the S1 ventilator for 5 hours, and compare to conventional ventilation.

DETAILED DESCRIPTION:
Research Design and Methods

Aim: To demonstrate the safety, feasibility and efficacy of delivering ventilator support in intubated children during the weaning phase with S1 ventilator using CO2 removal and O2 delivery explicit computerized protocol (ECP).

Hypothesis: The computerized explicit protocol implemented in S1 ventilator will better maintain children in a normal oxygen saturation, respiratory rate and ETPCO2 range during the weaning phase when compared to usual care.

Eligible patients: All critically ill children will be considered eligible for this research project if they fulfill all the following criteria :

* The patients should be PICU-hospitalized
* Child under mechanical ventilation with an endotracheal tube for at least 12 hours, as estimated by the attending intensivist.
* Child below 18 years of age, with a body weight ≥ 3 kg.

Screening of eligible patients: The attending Pediatric Intensivist and a Research Nurse will check for candidates on a daily basis in the pediatric intensive care unit (PICU) of Sainte-Justine Hospital (HSJ). An eligibility screening log, documenting the subject's fulfillment of the entry criteria, will be completed for all eligible patients considered for the study, regardless of their subsequent inclusion or exclusion status ("Bookkeeping"). Consent will be solicited from parents or legal guardians if a patient fulfils eligibility criteria and presents no exclusion criteria.

Inclusion and exclusion Criteria (see below)

Baseline data:

All subjects included into this study will undergo routine examination upon admission to the hospital. These examinations include physical, medical/medication history (on the last year for medical history and the last 3 months for medication history (if available)), vital signs, radiologic data and laboratory tests. Assessment of these data will occur in potential candidates within 24 hours of their hospitalization. BMI (Body Mass Index) will be derived from the subjects' height and weight. PIM 2 and PELOD scores will be computed (the PIM 2 score is a mortality risk score for children, and the PELOD score is a scale estimating the severity of cases of multiple organ).

Measurements:

Set and measured ventilatory parameters, SpO2 and ETPCO2 will be stored in the S1 ventilator. SpO2 will be measured via pulse oximetry placed on infant's extremities (in addition to usual monitoring) during the 5 hours of the study. End Tidal PCO2 measurements will also be made via probe placed on the Y piece of the respirator circuit (usual practice) during the 5 hours of the study.

General protocol sequence:

* All patients in the PICU at HSJ screened daily for eligibility
* Eligible cases reviewed with attending team and study team
* Informed consent obtained from parents or guardian
* Pressure support test A pre-inclusion test (pressure support test) with a level of pressure support of ± 5 cmH2O of the previous level of positive inspiratroy pressure in the controlled mode (PCV for instance), but no greater than 30 cmH2O (pressure-support level plus positive end-expiratory pressure), is performed to evaluate if the patient's is ready to be weaned. The test could be stopped before 30 minutes if the patient showed evidence of respiratory distress (respiratory rate > 40 breaths per minute and FiO2 > 60% in order to obtain pulse oxymetry ≥ 95%) or apnea. The test will be performed again the day after if he still reach inclusion/exclusion criteria. The test is considered positive when, after 30 minutes, the patient remained clinically stable with a respiratory rate between 10 and 40 breaths per minute and an expiratory tidal volume higher than 6 ml per kilogram of body weight within the authorized pressure-support range, with pulse oxymetry no lower than 95 percent when the fraction of inspired oxygen was no greater than 60 percent. When the pressure-support test is positive, the patient is included in the study.
* Data registered 1 hour in pressure support mode with the ventilator and settings of the pre-inclusion test.
* Ventilation is switched to S1 ventilator and the routine ventilator is kept in the patient room.
* Application of 3 hours with the S1 ventilator with the following initial settings:

At the study beginning, the S1 ventilator will be implemented and the settings used will be:

* ASV mode with % minute volume (MV) set as compared to the mean patient's MV measured during the 1 hour pressure support before
* PEEP: same as in conventional ventilation
* FIO2: same as in conventional ventilation After 1 hour, the CO2 removal ECP is started and 1 hour later, the O2 delivery ECP is started for 1 hour (figure 3).

  * Return to routine ventilator with the settings used at inclusion and registered during 1 hour A physician or respiratory therapist trained to use S1 ventilator will stay during the whole period (5 hours) next to the patient.

Monitoring during conventional ventilation after discontinuation of S1 ventilator (1 hour):

In order to compare S1 ventilator to conventional ventilation, monitoring will be continued with conventional settings on the usual ventilator for 1 hour. Following this, the study will be stopped and patient back to conventional ventilator unless attending physician decides to extubate the patient.

Protocol termination criteria: If the child demonstrates a sustained change in any of the following, the protocol will be terminated and the child ventilated with the previous conventional ventilation:

* Sustained decrease in SaO2 < 92% requiring increase in FIO2 > 60%
* ETPCO2 > ETPCO2 at S1 start requiring increase of positive inspiratory pressure > 25 cmH2O above PEEP,
* Sustained increase in heart rate > 180 bpm during 15 min,
* Sustained increase in respiratory rate > 60 bpm during 15 min,
* Uncontrolled agitation judged by the attending physician

Management of protocol termination episodes:

All protocol termination episodes will be analyzed by two pediatric intensivists non involved in the research project (François Proulx MD, France Gauvin MD). We do not expect any safety issue while performing this research project, but there is few experience with the S1 ventilator under study, which explain why we will so closely watch for any problem attributable to S1 ventilator.

Analysis and statistics Data will be described as n, mean, median, standard deviation, minimum and maximum for quantitative variables and frequencies for qualitative variables. The percentage of time in normal breathing range and normal saturation range will be compared between the last hour with S1 ventilator, and the first hour in conventional ventilation; and between the last hour with S1 ventilator and last hour in conventional ventilation 2 groups using a Wilcoxon's test.

ELIGIBILITY:
Inclusion Criteria:

An eligible subject will be considered for inclusion into this clinical trial if the attending physician is ready to begin weaning from mechanical ventilation and if the patient fulfils all the following inclusion criteria:

* The attending physician thinks that the patient will be able to breathe spontaneously or the patient is already breathing spontaneously.
* No vasopressor or inotropic medication, unless the patient is receiving some digitalin or small doses of dopamine or dobutamine (≤ 5 µg/kg/min)
* Slight or no endotracheal tube gas-leakage ((Vti - Vte)/Vti ≤ 20%)
* Mechanical ventilation with a plateau pressure ≤ 25 cmH2O over PEEP
* PEEP ≤ 8 cmH2O
* FiO2 ≤ 60% in order to obtain pulse oxymetry ≥ 95%
* PaCO2 < 70 mmHg on the last blood gases
* Extubation not expected the day of inclusion
* Gap between ETPCO2 and PCO2 < 7 mmHg on last blood gas.

Exclusion Criteria:

A patient will be excluded from this study a priori if he/she presents one or many of the following criteria:

* The patient fails the pressure-support test (this test is described below in the section entitled "Intervention").
* Invasive or non invasive mechanical ventilation at home or on hospital ward before PICU admission.
* Child with a tracheotomy
* Child with an history of mechanical ventilation > 2 months
* Contemplate withdrawing mechanical ventilation for palliative care
* Child with tracheobronchomalacia responsible for chronic respiratory failure
* Child with a severe neuromuscular disease prior to admission or acquired in the PICU and unable to generate a negative pressure of at least - 20 cmH20 during inspiration.
* Child with a "do not resuscitate order" and/or "do not reintubate order" is prescribed
* The child is still receiving some curare
* Cyanotic congenital heart disease with unrepaired or palliated right to left intracardiac shunt.
* Primary pulmonary hypertension.
* Child not expected to survive within a week, according to the attending intensivist
* Brain death or suspected brain death
* Morbid obesity defined by a body mass index (Actual Body Weight/T² > 40)
* Pregnant patient
* Parents or tutors do not agree to sign the consent form
* S1 ventilator is not available
* SpO2 monitoring not available (no plethysmographic curve) or not reliable
* EtCO2 not available (no capnogram) or no reliable (see above "gap")

Ages: 1 Hour to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time in acceptable breathing range | one hour
  Normal breathing range is defined as:
  In children age ≤ 2 years old: RR between 15 and 60 bpm and a tidal volume above 5 ml/kg of ideal body weight.
  In children > 2 years old: RR between 10 and 50 bpm and a tidal volume above 5 ml/kg of ideal body weight.

SECONDARY OUTCOMES:
Time in acceptable saturation range | 1 hour
  Acceptable saturation range is an SpO2 between 92% and 98%

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Jouvet, MD PhD, Principal Investigator — Sainte-Justine Hospital - University of Montreal
Locations (1):
- Sainte-Justine Hospital - University of Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Santschi M, Gauvin F, Hatzakis G, Lacroix J, Jouvet P. Acceptable respiratory physiologic limits for children during weaning from mechanical ventilation. Intensive Care Med. 2007 Feb;33(2):319-25. doi: 10.1007/s00134-006-0414-0. Epub 2006 Oct 25. PMID 17063358
- [Background] Jouvet P, Farges C, Hatzakis G, Monir A, Lesage F, Dupic L, Brochard L, Hubert P. Weaning children from mechanical ventilation with a computer-driven system (closed-loop protocol): a pilot study. Pediatr Crit Care Med. 2007 Sep;8(5):425-32. doi: 10.1097/01.PCC.0000282157.77811.F9. PMID 17693913
- [Background] Arnal JM, Wysocki M, Nafati C, Donati S, Granier I, Corno G, Durand-Gasselin J. Automatic selection of breathing pattern using adaptive support ventilation. Intensive Care Med. 2008 Jan;34(1):75-81. doi: 10.1007/s00134-007-0847-0. Epub 2007 Sep 11. PMID 17846747
- [Background] Sulemanji D, Marchese A, Garbarini P, Wysocki M, Kacmarek RM. Adaptive support ventilation: an appropriate mechanical ventilation strategy for acute respiratory distress syndrome? Anesthesiology. 2009 Oct;111(4):863-70. doi: 10.1097/ALN.0b013e3181b55f8f. PMID 19741490
- [Derived] Jouvet P, Eddington A, Payen V, Bordessoule A, Emeriaud G, Gasco RL, Wysocki M. A pilot prospective study on closed loop controlled ventilation and oxygenation in ventilated children during the weaning phase. Crit Care. 2012 May 16;16(3):R85. doi: 10.1186/cc11343. PMID 22591622